CLINICAL TRIAL: NCT07289113
Title: Personalized PEEP Titration Guided by Electrical Impedance Tomography in Patients Undergoing Laparoscopic Surgery: A Randomized Controlled Trial - The PEaRL Study
Brief Title: PEEP Titration Guided by Electrical Impedance Tomography in Laparoscopic Surgery The PEaRL Study
Acronym: PEaRL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Tommaso Fossali, Medical Doctor, head of the anesthesiologists, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CET 341-2025
Record Dates: First submitted 2025-11-19; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Electrical Impedance Tomography
Keywords: PEEP; Electrical Impedance Tomography; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard PEEP (No Intervention): PEEP value will be decided by clinician
- EIT PEEP (Experimental): PEEP value will be set after a PEEP trial performed with EIT machine
  Interventions: Device: A PEEP trial performed with the PulmoVista® 500 (Dräger, Lübeck, Germany) is a procedure designed to identify the optimal level of positive end-expiratory pressure

INTERVENTIONS:
Device: A PEEP trial performed with the PulmoVista® 500 (Dräger, Lübeck, Germany) is a procedure designed to identify the optimal level of positive end-expiratory pressure — During the trial, stepwise adjustments of PEEP are made while EIT provides real-time, bedside visualization of ventilation distribution across different lung regions. Typically, the protocol involves a recruitment maneuver followed by incremental and/or decremental PEEP steps (for example, in 2-3 cmH₂O intervals). At each step, EIT measures changes in regional impedance, which reflect variations in local lung aeration and ventilation.
  By analyzing these parameters, clinicians can determine the individualized "best PEEP", defined as the point at which alveolar collapse is minimized without causing significant overdistension. The optimal PEEP is then set for subsequent ventilation management.
  Arms: EIT PEEP

SUMMARY:
Background:

Laparoscopic surgery has gained widespread adoption due to its minimally invasive nature, offering advantages such as reduced postoperative pain, shorter hospitalization, and faster functional recovery compared with traditional open surgery. Nevertheless, postoperative respiratory complications remain a major source of morbidity. Factors such as general anesthesia, the Trendelenburg position, and CO₂ pneumoperitoneum can impair respiratory mechanics, reduce total lung capacity, and promote atelectasis, leading to compromised gas exchange.

Rationale:

Positive end-expiratory pressure (PEEP) is routinely applied to prevent alveolar collapse and improve oxygenation during mechanical ventilation. However, the use of standardized, non-individualized PEEP levels may be suboptimal, as inappropriate settings can cause alveolar overdistension or persistent collapse. Personalized PEEP titration, tailored to patient-specific lung mechanics, has recently emerged as a promising strategy to minimize ventilator-induced lung injury (VILI).

Methods and Tools:

Electrical Impedance Tomography (EIT) is a non-invasive, bedside monitoring technique that enables real-time assessment of regional lung ventilation. By evaluating ventilated and non-ventilated lung areas, EIT can guide PEEP optimization and support individualized ventilatory management. Recent studies suggest that EIT-guided PEEP titration improves respiratory parameters and reduces atelectasis in patients undergoing major surgery.

Objective:

The present study aims to evaluate the efficacy of EIT-guided PEEP personalization in patients undergoing laparoscopic and robotic surgery. Primary endpoints include improvements in regional ventilation, respiratory system compliance, and intraoperative gas exchange, as well as postoperative pulmonary function.

DETAILED DESCRIPTION:
Laparoscopic surgery has become an increasingly widespread surgical approach due to its minimally invasive nature, which allows for reduced postoperative pain, shorter hospital stays, and faster functional recovery compared to traditional open surgery. However, despite these advantages, laparoscopic procedures are not free from postoperative respiratory complications, which remain among the leading causes of postoperative morbidity. The combination of general anesthesia, the Trendelenburg position, and insufflation of CO₂ into the abdominal cavity can alter respiratory mechanics, reduce total lung capacity, and promote the development of atelectatic areas, resulting in impaired gas exchange (1-2).

Positive end-expiratory pressure (PEEP) is a widely used strategy to prevent alveolar collapse and improve oxygenation during mechanical ventilation. Nevertheless, the application of a standardized, non-individualized PEEP level may not be optimal for all patients, and an inappropriate PEEP setting may lead to alveolar overdistension or persistence of collapsed areas (3). Recently, personalized PEEP titration has gained attention as a method to tailor ventilation settings to individual patient characteristics, thereby minimizing the risk of ventilator-induced lung injury (VILI) (4).

Electrical Impedance Tomography (EIT) is a non-invasive, bedside imaging technique that enables real-time assessment of the regional distribution of pulmonary ventilation. EIT allows continuous monitoring of the effects of PEEP on both ventilated and non-ventilated lung regions and can guide the optimization of individualized PEEP levels to improve ventilation distribution and reduce the risk of respiratory complications (5-6). Recent studies have shown that the use of EIT-guided PEEP personalization in patients undergoing major surgery can improve respiratory parameters and reduce atelectasis formation (7-8). Specifically, EIT enables the performance of a PEEP trial, during which the device identifies areas of alveolar overdistension or collapse in response to PEEP changes, thereby guiding personalized ventilatory settings.

However, the application of this technique in the context of laparoscopic surgery remains limited. This study aims to evaluate the effectiveness of EIT-guided PEEP personalization in patients undergoing laparoscopic and robotic procedures, with the goal of improving regional ventilation, respiratory system compliance, and intraoperative gas exchange, as well as postoperative pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for laparoscopic abdominal surgery
* informed consent signed

Exclusion Criteria:

* COPD
* Acute respiratory failure
* Hemodynamic instability
* Pregnancy
* Contraindications for EIT device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Static respiratory system compliance | - Baseline (after anesthesia induction) - T1 (After Trendelemburg position and induction of pneumoperitoneum) - T2 (After PEEP trial) - T3 (90 minutes after PEEP trial) - T4 (180 minutes after PEEP trial) - T5 (Before end of anesthesia)
  Respiratory system compliance is equivalent to tidal volume divided by the diiference between plateau and PEEP pressure. Unit of measurement is cmH2O/mL

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Fossali, MD, Principal Investigator — ASST Fatebenefratelli Sacco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ma X, Fu Y, Piao X, De Santis Santiago RR, Ma L, Guo Y, Fu Q, Mi W, Berra L, Zhang C. Individualised positive end-expiratory pressure titrated intra-operatively by electrical impedance tomography optimises pulmonary mechanics and reduces postoperative atelectasis: A randomised controlled trial. Eur J Anaesthesiol. 2023 Nov 1;40(11):805-816. doi: 10.1097/EJA.0000000000001901. Epub 2023 Sep 13. PMID 37789753
- [Result] Rauseo M, Spadaro S, Mirabella L, Cotoia A, Laforgia D, Gaudino G, Vinella F, Ferrara G, Gattullo A, Tullo L, Cinnella G. Electrical Impedance Tomography during Abdominal Laparoscopic Surgery: A Physiological Pilot Study. J Clin Med. 2023 Dec 1;12(23):7467. doi: 10.3390/jcm12237467. PMID 38068519
- [Result] Jiang L, Deng Y, Xu F, Qiao S, Wang C. Individualized PEEP guided by EIT in patients undergoing general anesthesia: A systematic review and meta-analysis. J Clin Anesth. 2024 Jun;94:111397. doi: 10.1016/j.jclinane.2024.111397. Epub 2024 Jan 25. PMID 38278058
- [Result] Pavlovsky B, Desprez C, Richard JC, Fage N, Lesimple A, Chean D, Courtais A, Mauri T, Mercat A, Beloncle F. Bedside personalized methods based on electrical impedance tomography or respiratory mechanics to set PEEP in ARDS and recruitment-to-inflation ratio: a physiologic study. Ann Intensive Care. 2024 Jan 5;14(1):1. doi: 10.1186/s13613-023-01228-4. PMID 38180544
- [Result] Gao Y, He H, Chi Y, Frerichs I, Long Y, Zhao Z. Electrical impedance tomography guided positive end-expiratory pressure titration in critically ill and surgical adult patients: a systematic review and meta-analysis. BMC Pulm Med. 2024 Nov 23;24(1):582. doi: 10.1186/s12890-024-03394-y. PMID 39580405
- [Result] Chen L, Yu K, Yang J, Han X, Liu L, Li T, Miao H. Electrical impedance tomography-guided positive end-expiratory pressure titration for perioperative oxygenation and postoperative pulmonary complications: A systematic review and meta-analysis. Medicine (Baltimore). 2024 Dec 27;103(52):e40357. doi: 10.1097/MD.0000000000040357. PMID 39969340
- [Result] Scaramuzzo G, Priani P, Ferrara P, Verri M, Montanaro F, La Rosa R, Cammarota G, Volta CA, Spadaro S. Longitudinal changes of electrical impedance tomography-based best PEEP in obese patients undergoing laparoscopic surgery: A prospective physiological study. Anaesth Crit Care Pain Med. 2025 Sep;44(5):101569. doi: 10.1016/j.accpm.2025.101569. Epub 2025 Jun 13. PMID 40518045